CLINICAL TRIAL: NCT01680939
Title: Investigating the Safety of Morphine and Ibuprofen in Children Post-adenotonsillectomy for Obstructive Sleep Apnea
Brief Title: Investigating the Safety of Post-surgical Analgesics in Children With Obstructive Sleep Apnea
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: The Hospital for Sick Children (Other); University of Western Ontario, Canada (Other)
Responsible Party: Principal Investigator, Doron Sommer, MD, Hamilton Health Sciences Corporation
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSAS-HHSC2012
Record Dates: First submitted 2012-09-04; First posted 2012-09-07 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: Pediatric Obstructive Sleep Apnea Syndrome
Keywords: Pediatrics; Obstructive Sleep Apnea; Adenotonsillectomy; Analgesia
MeSH Terms: conditions — Sleep Apnea, Obstructive; Agnosia | interventions — Morphine; Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Morphine (Experimental): Receives morphine for post-surgical pain
  Interventions: Drug: Morphine
- Ibuprofen (Experimental): Receives ibuprofen for post-surgical pain
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Morphine — 0.2-0.5 mg/kg PO q4h
  Arms: Morphine
Drug: Ibuprofen — 10mg/kg PO q6hrs
  Arms: Ibuprofen

SUMMARY:
Every year thousands of young children with obstructive sleep apnea undergo surgery which requires them to be prescribed pain medication. The current standard in North America is administration of opioids, mainly codeine or morphine; however in many areas of the world including Canada, nonsteroidal anti-inflammatory medications such as ibuprofen are used. Some North American surgeons are uncertain regarding the potential of ibuprofen to increase bleeding following surgery. The results of research studies have been inconclusive overall. Due to recent codeine fatalities in children following adenotonsillectomy, codeine has been removed from the formulary at many Pediatric institutions. Some surgeons have begun to use oral morphine as an alternate to codeine, which necessitates the need to find safe alternative analgesics in this treatment group.

The primary objectives of this study is to assess the safety(1) and efficacy (2) of morphine and ibuprofen in children with sleep apnea.

An interim analysis will be conducted after recruitment of 70 patients, to monitor both safety and efficacy

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with OSAS,
* scheduled for tonsillectomy plus/minus adenoid removal at MUMC,
* between the ages of 1-10years

Exclusion Criteria:

* contraindications to analgesia,
* asthma,
* has had previous adenotonsillectomy, or
* any craniofacial,
* neuromuscular or cardiac conditions

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Safety | 1.5 years
  Safety will be assessed by comparing changes in respiratory parameters (oxygen saturation and the number of apnea events per night) following adenotonsillectomy.

SECONDARY OUTCOMES:
Effectiveness | 1.5 years
  Analgesic effectiveness between treatment groups will be assessed using the visual analog scale and the objective pain scale
Risk Factors | 1.5 years
  Age, BMI, OSA severity and genetic factors will be compared between treatment groups. Furthermore, these factors will be isolated to determine any correlation exists with respiratory parameter improvement in all enrolled patients.

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University Medical Centre, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Kelly LE, Sommer DD, Ramakrishna J, Hoffbauer S, Arbab-Tafti S, Reid D, Maclean J, Koren G. Morphine or Ibuprofen for post-tonsillectomy analgesia: a randomized trial. Pediatrics. 2015 Feb;135(2):307-13. doi: 10.1542/peds.2014-1906. PMID 25624387